CLINICAL TRIAL: NCT00467831
Title: Pilot Study of a Multi-Drug Regimen for Severe Pulmonary Fibrosis in Hermansky-Pudlak Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070132; 07-HG-0132 (Other: NHGRI IRB)
Record Dates: First submitted 2007-04-28; First posted 2007-05-01 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Hermansky-Pudlak Syndrome (HPS); Pulmonary Fibrosis; Oculocutaneous Albinism; Platelet Storage Pool Deficiency; Metabolic Disease
Keywords: Restrictive Lung Disease; Pulmonary Fibrosis; Albinism; Platelet Storage Pool Deficiency; Metabolic Disease; Hermansky-Pudlak Syndrome; HPS; Lung Disease
MeSH Terms: conditions — Hermanski-Pudlak Syndrome; Pulmonary Fibrosis; Albinism, Oculocutaneous; Platelet Storage Pool Deficiency; Metabolic Diseases; Albinism; Lung Diseases | interventions — Losartan; zileuton; Acetylcysteine; Pravastatin; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi-Drug Regimen (Experimental): Losartan, 25 mg by mouth every night at bedtime; Zileuton, 1200 mg by mouth twice daily; N-acetylcysteine, 600 mg by mouth three times daily; Pravastatin, 20 mg by mouth every night at bedtime; Erythromycin, 333 mg by mouth three times daily.
  Interventions: Drug: Losartan; Drug: Zileuton; Drug: N-Acetylcysteine; Drug: Pravastatin; Drug: Erythromycin

INTERVENTIONS:
Drug: Losartan — Losartan potassium tablet, 25 mg by mouth every night at bedtime.
  Other Names: Cozaar
Drug: Zileuton — Zileuton tablet, 1200 mg by mouth twice daily.
  Other Names: Zyflo
Drug: N-Acetylcysteine — N-acetylcysteine solution, 600 mg by mouth three times daily.
  Other Names: acetylcysteine
Drug: Pravastatin — Pravastatin sodium tablet, 20 mg by mouth every night at bedtime.
  Other Names: Pravachol
Drug: Erythromycin — Erythromycin tablet, 333 mg by mouth three times daily.
  Other Names: E-mycin; Ery-tab

SUMMARY:
This study will examine whether five drugs (pravastatin, Losartan, Zileuton, N-acetylcysteine and erythromycin) used together can slow the course of pulmonary fibrosis (scarring of the lung tissue) in patients with Hermansky-Pudlak Syndrome (HPS). Patients with this disease have decreased skin color (albinism), bleeding problems, and sometimes colon problems. Two of the known types of Hermansky Pudlak syndrome, type 1 and type 4, are at high risk of pulmonary fibrosis between the ages of 30 and 50.

Patients 18 to 70 years of age who have Hermansky-Pudlak Syndrome with a serious loss of lung function due to pulmonary fibrosis may be eligible for this study.

Participants begin taking pravastatin on study day 2 and start a new drug every 3 days. Patients who experience no problems with the medicines return home and continue on the drugs for the next 2 years. They return to the NIH Clinical Center every 3 months for a medical history, physical examination, and blood, urine and lung function tests. CT and bone density scans are done every year. The study may continue for up to 3 years.

DETAILED DESCRIPTION:
Hermansky-Pudlak Syndrome (HPS) is a rare autosomal recessive disease consisting of oculocutaneous albinism and a platelet storage pool defect. The most serious complication of this disorder, pulmonary fibrosis, occurs only in genetic subtypes HPS-1 and HPS-4 and is generally fatal in the fourth or fifth decade. HPS-1 is very common in northwest Puerto Rico. There is no effective treatment for the pulmonary disease of HPS (HPS-PF), which resembles idiopathic pulmonary fibrosis (IPF). A preliminary study of the antifibrotic drug, pirfenidone, gave promising results for mild to moderate HPS-PF, but not for severe pulmonary fibrosis. A second study is currently addressing only mild to moderate HPS-PF. Other drugs, studied in IPF as single agents, have some efficacy for mild to moderate disease, but none has had a major effect on mortality. Recently, a call has been made for consideration of multi-drug therapy (i.e., an oncologic approach) for severe pulmonary fibrosis. Based upon positive responses from companies producing relevant drugs, we propose a multi-drug trial using five agents: Losartan, Zileuton, a generic statin (Pravastatin), generic N-acetylcysteine, and generic Erythromycin. Participants with severe pulmonary fibrosis will be drawn largely from the Puerto Rican population. Eligibility will require a molecular diagnosis of HPS-1 or HPS-4, radiographic evidence of interstitial lung disease, persistent pulmonary function testing less than or equal to 45% of predicted after bronchodilation, and absence of other causes of lung dysfunction. Participants will be admitted to the NIH Clinical Center for a 21-day admission to establish baseline function and to begin medication therapy. Follow-up admissions (3 days) will occur every 3 months. The primary outcome parameter will be survival at 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this protocol, participants must:

* Have a molecular diagnosis of HPS-1 or HPS-4
* Be 18-70 years of age
* Have the expectation to live more than 3 months, i.e., an FVC greater than or equal to 30% of predicted
* Have evidence of severe pulmonary fibrosis, i.e.:

  1. A FVC less than or equal to 45% of predicted
  2. Reduced exercise tolerance lasting longer than 1 week on the Dyspnea Perception Scale
  3. No evidence of improvement in pulmonary fibrosis within the past year, as defined by an FVC increase of 10% or a DLco increase of 15%.
* Be available, willing, and able to come to the NIH Clinical Center for admission every 3 months.

EXCLUSION CRITERIA:

* An explanation for interstitial lung disease other than HPS, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, cancer
* Pregnancy or lactation
* History of ethanol abuse or recreational drug use in the past two years
* History of human immunodeficiency virus (HIV) or chronic viral hepatitis infection
* Chronic use of high-dose steroids (greater than 10 mg prednisone/day) intended for ongoing treatment of their interstitial lung disease
* Use of any of the following within 28 days of enrollment: investigational therapy, cytotoxic/immunosuppressive agents other than corticosteroids, including but not limited to azathioprine, cyclosphosphamide, methotrexate, cyclosporine, colchicine, interferon gamma-1b, bosentan;
* Any severe medical complication including but not be limited to uncontrolled seizures, repeated transient ischemic attacks, severe ataxia, uncontrolled migraine headaches, diplopia, repeated episodes of syncope, an untreated psychiatric disorder, recent myocardial infarction (past 6 months), unstable angina, clinically relevant and untreated arrhythmias, uncontrolled hypotension or hypertension (systolic blood pressure less than 80 or greater than 180 mm Hg), myocarditis, severe congestive left sided heart failure, hepatomegaly not due to right heart failure, renal glomerular impairment (creatinine clearance less than 35 ml/min/1.73 m(2)), pancreatitis, toxic thyroiditis, life-threatening malignancy;NOTE: right sided heart failure due to pulmonary hypertension as a result of pulmonary fibrosis will not be considered an exclusion criteria.
* Significant laboratory abnormalities, including but not limited to serum potassium less than 3.0 or greater than 5.4 mEq/L, SGPT greater than 100 U/L, CK greater than 700 U/L, hemoglobin less than 9.0 g/dL, platelets less than 70 k/mm(3), leukocyte count less than 2.0 k/microL;
* For women of child-bearing age, failure to have an effective method of birth control. Oral contraceptives will be considered inadequate without a second method due to risk of reduced efficacy of BCP while taking Zileuton.
* Severe psychiatric disease untreated. Inability to give informed consent after reading or having the consent read to the participant in their native language. Any concern that there is a therapeutic misconception will be evaluated by genetic counselor and/or appropriate mental health professionals prior to acceptance into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Markello, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Witkop CJ, Nunez Babcock M, Rao GH, Gaudier F, Summers CG, Shanahan F, Harmon KR, Townsend D, Sedano HO, King RA, et al. Albinism and Hermansky-Pudlak syndrome in Puerto Rico. Bol Asoc Med P R. 1990 Aug;82(8):333-9. PMID 2261023
- [Background] HERMANSKY F, PUDLAK P. Albinism associated with hemorrhagic diathesis and unusual pigmented reticular cells in the bone marrow: report of two cases with histochemical studies. Blood. 1959 Feb;14(2):162-9. No abstract available. PMID 13618373
- [Background] Huizing M, Gahl WA. Disorders of vesicles of lysosomal lineage: the Hermansky-Pudlak syndromes. Curr Mol Med. 2002 Aug;2(5):451-67. doi: 10.2174/1566524023362357. PMID 12125811
- [Background] Introne WJ, Huizing M, Malicdan MCV, O'Brien KJ, Gahl WA. Hermansky-Pudlak Syndrome. 2000 Jul 24 [updated 2023 May 25]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1287/ PMID 20301464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from April 2007 to November 2012 at the NIH Clinical Center.
Groups:
- Multi-Drug Regimen: Losartan, 25 mg by mouth every night at bedtime; Zileuton, 1200 mg by mouth twice daily; N-acetylcysteine, 600 mg by mouth three times daily; Pravastatin, 20 mg by mouth every night at bedtime; Erythromycin, 333 mg by mouth three times daily.
  Erythromycin : Erythromycin tablet, 333 mg by mouth three times daily.
  Losartan : Losartan potassium tablet, 25 mg by mouth every night at bedtime.
  Zileuton : Zileuton tablet, 1200 mg by mouth twice daily.
  N-Acetylcysteine : N-acetylcysteine solution, 600 mg by mouth three times daily.
  Pravastatin : Pravastatin sodium tablet, 20 mg by mouth every night at bedtime.
Period: Overall Study
Arm/Group | Multi-Drug Regimen
Started | 3
Completed | 0
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Multi-Drug Regimen
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Survival at 2 Years
Description: The number of subjects surviving after 24 months on study.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Multi-Drug Regimen
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: Overall study: 24 months
Arm/Group | Multi-Drug Regimen
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-Drug Regimen (N=3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — respiratory failure due to end stage lung disease resulting in death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-Drug Regimen (N=3)
elevated liver enzyme levels (Hepatobiliary disorders) | 2 (2)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
anemia (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated because enrollment was too low. The results shown are not statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes